CLINICAL TRIAL: NCT01483183
Title: A Multi-center, Parallel-group, Double-blind, Placebo-controlled, Randomized, Ascending Dose Trial to Determine the Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous Infusions of OPC-108459 Administered to Subjects With Paroxysmal and Persistent Atrial Fibrillation
Brief Title: Ascending Dose Study of OPC-108459 Intravenous Infusions in Patients With Paroxysmal and Persistent Atrial Fibrillation
Acronym: CADENCE 215
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment Difficulty
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 269-11-215
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Paroxysmal Atrial fibrillation; Persistent Atrial fibrillation; A-fib
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Persistent or Paroxysmal AF Part 1: OPC-108459 (Experimental): To safely meet each of the following Cmax targets: 1.0-10.0 µg/mL. There will be 9 cohorts in all: 1.0, 1.6, 2.4, 3.6, 5.4, 7.0, 8.0, 9.0, and 10.0.
  Interventions: Drug: OPC-108459
- Persistent or Paroxysmal AF Part 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Persistent or Paroxysmal AF Part 2: OPC-108459 (Experimental): Single dose to safely meet target concentration from Part 1, if subject fails to convert to sinus rhythm within 10 minutes, second dose will be administered to achieve 25% increase when compared to first infusion
  Interventions: Drug: OPC-108459
- Placebo Part 2 (Placebo Comparator)
  Interventions: Drug: OPC-108459; Drug: Placebo

INTERVENTIONS:
Drug: OPC-108459 — Part 1: single dose OPC-108459, 10-minute constant rate IV infusion to achieve specified Cmax target
  Part 2: single dose OPC-108459, 10-minute constant rate IV infusion to achieve Cmax target concentration from Part 1; if failure to convert to sinus rhythm, second dose OPC-108459 administered, 10-minute constant rate IV infusion to achieve target concentration from Part 1
  Other Names: 269-11-215
  Arms: Persistent or Paroxysmal AF Part 1: OPC-108459; Persistent or Paroxysmal AF Part 2: OPC-108459; Placebo Part 2
Drug: Placebo — Placebo dose, 10-minute constant rate IV infusion
  Arms: Persistent or Paroxysmal AF Part 1: Placebo; Placebo Part 2

SUMMARY:
The purpose of Part 1 of this study is to determine the maximally tolerated dose of OPC-108459 in patients with paroxysmal and persistent atrial fibrillation (AF).

The purpose of Part 2 of this study is to determine potential efficacy of dose(s) of OPC-108459 for the treatment of paroxysmal and persistent atrial fibrillation.

DETAILED DESCRIPTION:
This trial will test the pharmacokinetic and pharmacodynamic characteristics of ascending doses of OPC-108459 in separate populations of paroxysmal and persistent AF subjects.

The trial will consist of two parts. Each part will evaluate two populations of subjects presenting for cardioversion in a hospital setting.

Cohorts of paroxysmal and persistent subjects may have their dose increased independently.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with paroxysmal atrial fibrillation (AF) (recent or new onset) or subjects with persistent AF at the time of randomization
* Subjects who are hemodynamically stable
* Subjects with a low risk of thromboembolic potential
* Subjects who are willing to comply with the reproductive precautions

Exclusion Criteria:

Subjects with:

* History of long QT syndrome, Torsade de Pointes or an uncorrected QT interval of > 450 ms
* History of myocardial infarction within 6 months of screening
* Acute coronary syndrome, angina or active myocardial ischemia diagnosed by ECG, or other imaging within 6 months of screening
* History of ventricular tachycardia, fibrillation, or resuscitated cardiac arrest
* History of clinically significant congenital heart disease
* Presence of severe aortic or mitral stenosis, aortic or mitral regurgitation, atrial septal defect, or other conditions leading to AF
* Diagnosis of heart failure NYHA Class II-IV or with an ejection fraction <40% (Part 1 only)
* Diagnosis of heart failure NYHA Class IV or NYHA I, II, or III with an ejection fraction <35% (Part 2 only)
* Concomitant treatment with class I or III anti-arrhythmics agents unless the medication was discontinued more than 5 half-lives before dosing
* History of seizures
* Diagnosis of atrial flutter
* Diagnosis of stroke, TIA (transient ischemic attack), or any transient neurological deficit within 1 year of screening or known carotid artery stenosis of >50%
* Cardiac surgery within 3 months of screening
* Bradycardia (< 50 bpm) or sick sinus syndrome, unless controlled by a pacemaker
* Current reversible cause of AF
* Wolff-Parkinson-White syndrome
* Any congenital abnormality, severe valve disease
* Subjects who have taken another investigational product within 30 days of dosing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (9):
  - Otsuka Investigational Site, Washington D.C., District of Columbia
  - Otsuka Investigational Site, Hollywood, Florida
  - Otsuka Investigational Site, Jacksonville, Florida
  - Otsuka Investigational Site, Sarasota, Florida
  - Otsuka Investigational Site, Lexington, Kentucky
  - Otsuka Investigational Site, New Orleans, Louisiana
  - Otsuka Investigational Site, Johnson City, New York
  - Otsuka Investigational Site, Germantown, Tennessee
  - Otsuka Investigational Site, Houston, Texas
- Germany (4):
  - Otsuka Investigational Site, Berlin
  - Otsuka Investigational Site, Hamburg
  - Otsuka Investigational Site, Leipzig
  - Otsuka Investigational Site, Pirna
- Italy (4):
  - Otsuka Investigational Site, San Fermo, Como
  - Otsuka Investigational Site, Ancona
  - Otsuka Investigational Site, Bologna
  - Otsuka Investigational Site, Cremona
- Netherlands (2):
  - Otsuka Investigational Site, Amsterdam
  - Otsuka Investigational Site, Groningen
- Spain (4):
  - Otsuka Investigational Site, Fuenlabrada, Madrid
  - Otsuka Investigational Site, Barcelona
  - Otsuka Investigational Site, Granada
  - Otsuka Investigational Site, Madrid
- Otsuka Investigational Site, Chertsey, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 40 participants at 10 trial sites in the following 3 countries: Germany, Spain, and the United States.
Pre-assignment Details: The trial consists of two parts (Part 1 and Part 2). Each part evaluates two populations of participants for cardioversion in a hospital setting; one diagnosed with paroxysmal atrial fibrillation (AF) and the second diagnosed with persistent AF. However, Part 2 was not conducted and therefore is not included in this document.
Groups:
- Paroxysmal AF - OPC-108459 0.26 mg/kg: Participants received a single dose of OPC-108459 0.26 milligram per kilogram (mg/kg), 10-minute constant rate intravenous (IV) infusion to achieve specified Cmax target.
- Paroxysmal AF - OPC-108459 0.40 mg/kg; Persistent AF - OPC-108459 0.40 mg/kg: Participants received a single dose of OPC-108459 0.40 mg/kg,10-minute constant rate IV infusion to achieve specified Cmax target.
- Paroxysmal AF - OPC-108459 1.00 mg/kg: Participants received a single dose of OPC-108459 1.00 mg/kg,10-minute constant rate IV infusion to achieve specified Cmax target.
- Paroxysmal AF - Placebo: Participants received placebo dose 10-minute constant rate IV infusion.
- Persistent AF - OPC-108459 0.26 mg/kg: Participants received a single dose of OPC-108459 0.26 mg/kg,10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - OPC-108459 0.60 mg/kg: Participants received a single dose of OPC-108459 0.60 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - OPC-108459 1.35 mg/kg: Participants received a single dose of OPC-108459 1.35 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - OPC-108459 1.55 mg/kg: Participants received a single dose of OPC-108459 1.55 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - Placebo: Participants received a single dose of placebo, 10-minute constant rate IV infusion.
Period: Overall Study
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo
Started | 4 | 1 | 5 | 3 | 4 | 4 | 6 | 4 | 4 | 5
Completed | 4 | 1 | 5 | 3 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Paroxysmal AF - OPC-108459 0.26 mg/kg: Participants had received a single dose of OPC-108459 0.26 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Paroxysmal AF - OPC-108459 0.40 mg/kg; Persistent AF - OPC-108459 0.40 mg/kg: Participants had received a single dose of OPC-108459 0.40 mg/kg,10-minute constant rate IV infusion to achieve specified Cmax target.
- Paroxysmal AF - OPC-108459 1.00 mg/kg: Participants had received a single dose of OPC-108459 1.00 mg/kg,10-minute constant rate IV infusion to achieve specified Cmax target.
- Paroxysmal AF - Placebo: Participants had received placebo dose 10-minute constant rate IV infusion.
- Persistent AF - OPC-108459 0.26 mg/kg: Participants had received a single dose of OPC-108459 0.26 mg/kg,10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - OPC-108459 0.60 mg/kg: Participants had received a single dose of OPC-108459 0.60 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - OPC-108459 1.35 mg/kg: Participants had received a single dose of OPC-108459 1.35 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - OPC-108459 1.55 mg/kg: Participants had received a single dose of OPC-108459 1.55 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
- Persistent AF - Placebo: Participants had received a single dose of placebo, 10-minute constant rate IV infusion.
- Total: Total of all reporting groups
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo | Total
Number analyzed (Participants) | 4 | 1 | 5 | 3 | 4 | 4 | 6 | 4 | 4 | 5 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (19.0) | 75.0 (0.0) | 68.4 (9.1) | 61.0 (14.1) | 65.0 (5.7) | 75.0 (10.1) | 63.5 (14.7) | 64.8 (12.9) | 64.3 (7.7) | 70.4 (8.8) | 66.6 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 11
  Male | 3 | 0 | 2 | 2 | 3 | 3 | 5 | 4 | 3 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum (Peak) Plasma Concentration (Cmax)
Description: OPC-108459 was administered as a 10-minute constant rate IV infusion. Blood samples were collected pre-dose (within 45 minutes of dosing), at the end of infusion and 0.5, 1, 2, 4, 8 and 24 hours post start of infusion.
Time Frame: 24 hours
Population: PK analysis dataset included all participants who had concentration time profiles consistent with proper intravenous infusion.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg
Number analyzed (Participants) | 4 | 1 | 4 | 4 | 3 | 3 | 3 | 4
μg/mL | 1.11 (0.358) | 1.49 (NA) — Due to only 1 participant with evaluable data. | 2.96 (0.787) | 1.45 (1.43) | 1.54 (0.538) | 1.62 (1.07) | NA (NA) — The data was not evaluable as the PK was collected from the same line as the infusion. Hence, there is no data available. | 5.14 (1.26)

2. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time 0 to Time of the Last Measurable Concentration (AUCτ)
Description: OPC-108459 was administered as a 10-minute constant rate IV infusion. Blood samples were collected pre-dose (within 45 minutes of dosing), at the end of infusion and 0.5, 1, 2, 4, 8 and 24 hours post infusion.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg∙h/mL
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg
Number analyzed (Participants) | 4 | 1 | 4 | 4 | 3 | 3 | 3 | 4
μg∙h/mL | 1.94 (0.834) | 1.25 (NA) — Due to only 1 participant with evaluable data. | 2.10 (0.318) | 1.28 (0.388) | 1.68 (0.650) | 1.51 (0.651) | 2.79 (0.990) | 4.38 (1.55)

3. Primary Outcome: Part 1:Maximal Change From Baseline in QT Interval Corrected for Heart Rate Using the Fridericia Formula (QTcF) Within 24 Hour Infusion
Description: 12-lead Holter monitors were placed on all participants within 45 minutes prior to dosing. Post dose measurements were made at 2, 4, 6, 8, 10, 20, 30, and 40 minutes and 1, 1.5, 2, 4, 6, 8, 12, 16, and 24 hours post-dose. To achieve consistent recording, Holter sampling will be recorded with the participant recumbent and at rest for at least 10 minutes prior to collection.
Time Frame: 24 hours
Population: Safety dataset included all participants who had received at least one dose of the trial medication.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Paroxysmal AF - OPC-108459 0.40 mg/kg: Participants had received a single dose of OPC-108459 0.40 mg/kg, 10-minute constant rate IV infusion to achieve specified Cmax target.
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo
Number analyzed (Participants) | 4 | 1 | 5 | 2 | 4 | 4 | 4 | 3 | 4 | 5
msec
  Increase | 15.0 (8.0) | NA (NA) — Due to only 1 participant with evaluable data. | 28.8 (12.0) | 11.5 (10.6) | 24.5 (21.4) | 24.0 (9.5) | 23.3 (20.2) | 19.7 (6.5) | 42.5 (29.0) | 27.4 (22.9)
  Decrease | -30.8 (7.8) | NA (NA) — Due to only 1 participant with evaluable data. | -18.2 (7.8) | -37.0 (8.5) | -15.3 (9.6) | -17.8 (14.1) | -23.0 (6.5) | -18.7 (16.5) | -13.3 (14.0) | -25.8 (8.5)

4. Primary Outcome: Part 1: Maximal Change From Baseline in Ventricular Rate Within 24 Hour Infusion
Description: as for outcome 3
Time Frame: 24 hours
Population: Safety dataset included all participants who had received at least one dose of the trial medication.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo
Number analyzed (Participants) | 4 | 1 | 5 | 2 | 4 | 4 | 4 | 3 | 4 | 5
beats/minute
  Increase | 22.3 (18.5) | NA (NA) — Due to only 1 participant with evaluable data. | 14.6 (5.0) | 15.5 (6.4) | 19.5 (9.1) | 18.5 (6.2) | 14.8 (13.1) | 28.0 (5.0) | 31.5 (15.6) | 26.0 (13.2)
  Decrease | -14.3 (6.6) | NA (NA) — Due to only 1 participant with evaluable data. | -29.8 (26.6) | -24.0 (1.4) | -6.8 (6.4) | -12.3 (3.3) | -19.8 (13.5) | -11.5 (3.5) | -8.3 (6.4) | -12.4 (6.4)

5. Primary Outcome: Part 1: Maximal Change From Baseline in Blood Pressure Within 24 Hour Infusion
Description: Maximum change from baseline in diastolic and systolic blood pressure(BP) collected during vital sign measurements in the 24-hour postdose interval. Participants must be hemodynamically stable defined as a screening systolic blood pressure between 90 to 160 mmHg, diastolic <100 mmHg. BP was measured after at least 3 minutes in the supine position. BP was measured at predose (within 45 minutes of dosing); 3 and 7 minutes and approximately 1, 4, 8, 12, and 24 hours.
Time Frame: 24 hours
Population: Safety dataset included all participants who had received at least one dose of the trial medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo
Number analyzed (Participants) | 4 | 1 | 5 | 3 | 4 | 4 | 4 | 4 | 4 | 5
mmHg
  Diastolic BP Supine (Decrease) | -13.8 (11.4) | NA (NA) — Due to only 1 participant with evaluable data. | -13.4 (8.7) | -25.7 (18.3) | -13.5 (15.3) | -5.0 (4.2) | -14.5 (9.3) | -18.7 (24.6) | -19.0 (6.2) | -10.8 (5.5)
  Diastolic BP Supine (Increase) | 4.3 (2.5) | 26.0 (NA) — Due to only 1 participant with evaluable data. | 18.6 (25.1) | 8.0 (11.3) | 5.3 (5.1) | 5.0 (2.6) | 1.7 (0.6) | 9.8 (7.9) | 21.0 (6.7) | 10.2 (6.7)
  Systolic BP Supine (Decrease) | -11.3 (6.4) | NA (NA) — Due to only 1 participant with evaluable data. | -20.8 (14.1) | -18.3 (18.6) | -7.8 (5.7) | -3.0 (1.4) | -9.0 (6.2) | -17.3 (13.7) | -24.5 (10.5) | -23.0 (15.1)
  Systolic BP Supine (Increase) | 14.3 (10.4) | 42.0 (NA) — Due to only 1 participant with evaluable data. | 16.6 (11.9) | 14.3 (23.1) | 7.5 (8.4) | 11.3 (8.2) | 8.5 (7.5) | 21.7 (6.4) | 15.0 (6.4) | 12.1 (8.6)

6. Primary Outcome: Part 2/1 Infusion: Cmax
Description: The trial was terminated after Part 1 enrollment completed. All analyses described in this document were performed on Part 1 data. However, Part 2 was not conducted and therefore is not included in this document.
Time Frame: 24 hours
Reporting Status: Not Posted

7. Primary Outcome: Part 2/2 Infusions: Cmax
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

8. Primary Outcome: Part 2/1 Infusion: AUCt
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

9. Primary Outcome: Part 2/2 Infusions: AUCt
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

10. Primary Outcome: Part 2: QTcF
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

11. Primary Outcome: Part 2: Ventricular Rate
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

12. Primary Outcome: Part 2: Diastolic and Systolic Blood Pressure
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

13. Primary Outcome: Part 2: Percentage of Subjects With Normal Sinus Rhythm (NSR)
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

14. Secondary Outcome: Part 1: Percentage of Participants With NSR
Description: Percent of participants with NSR, defined as NSR for at least 1 minute within 30 minutes of the end of OPC-108459 infusion.
Time Frame: 30 minutes
Population: Safety dataset included all participants who had received at least one dose of the trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo
Number analyzed (Participants) | 4 | 1 | 5 | 3 | 4 | 4 | 4 | 4 | 4 | 5
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Part 2: Time to NSR
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

16. Secondary Outcome: Part 2: Duration of NSR
Description: as for outcome 6
Time Frame: 24 hours
Reporting Status: Not Posted

17. Secondary Outcome: Part 2: Duration of NSR
Description: as for outcome 6
Time Frame: 168 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent throughout the 8-day study until the final follow-up phone call Day 31 (+2) days post dose.
Arm/Group | Paroxysmal AF - OPC-108459 0.26 mg/kg | Paroxysmal AF - OPC-108459 0.40 mg/kg | Paroxysmal AF - OPC-108459 1.00 mg/kg | Paroxysmal AF - Placebo | Persistent AF - OPC-108459 0.26 mg/kg | Persistent AF - OPC-108459 0.40 mg/kg | Persistent AF - OPC-108459 0.60 mg/kg | Persistent AF - OPC-108459 1.35 mg/kg | Persistent AF - OPC-108459 1.55 mg/kg | Persistent AF - Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/5 | 1/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 1/5
Other Adverse Events (participants affected / at risk) | 1/4 | 1/1 | 2/5 | 0/3 | 0/4 | 1/4 | 0/4 | 1/4 | 1/4 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paroxysmal AF - OPC-108459 0.26 mg/kg (N=4) | Paroxysmal AF - OPC-108459 0.40 mg/kg (N=1) | Paroxysmal AF - OPC-108459 1.00 mg/kg (N=5) | Paroxysmal AF - Placebo (N=3) | Persistent AF - OPC-108459 0.26 mg/kg (N=4) | Persistent AF - OPC-108459 0.40 mg/kg (N=4) | Persistent AF - OPC-108459 0.60 mg/kg (N=4) | Persistent AF - OPC-108459 1.35 mg/kg (N=4) | Persistent AF - OPC-108459 1.55 mg/kg (N=4) | Persistent AF - Placebo (N=5)
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paroxysmal AF - OPC-108459 0.26 mg/kg (N=4) | Paroxysmal AF - OPC-108459 0.40 mg/kg (N=1) | Paroxysmal AF - OPC-108459 1.00 mg/kg (N=5) | Paroxysmal AF - Placebo (N=3) | Persistent AF - OPC-108459 0.26 mg/kg (N=4) | Persistent AF - OPC-108459 0.40 mg/kg (N=4) | Persistent AF - OPC-108459 0.60 mg/kg (N=4) | Persistent AF - OPC-108459 1.35 mg/kg (N=4) | Persistent AF - OPC-108459 1.55 mg/kg (N=4) | Persistent AF - Placebo (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The trial was terminated after Part 1 enrollment completed. It did not progress due to many factors including slow enrollment, limited site activity in pre-screening, absence of reproducible efficacy signal and increased costs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.